CLINICAL TRIAL: NCT00346164
Title: Risk-Based Treatment for Non-Rhabdomyosarcoma Soft Tissue Sarcomas (NRSTS) in Patients Under 30 Years of Age
Brief Title: Observation, Radiation Therapy, Combination Chemotherapy, and/or Surgery in Treating Young Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST0332; NCI-2009-00426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST0332 (Other: Children's Oncology Group); CDR0000483702 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-06

CONDITIONS: Adult Alveolar Soft-part Sarcoma; Adult Angiosarcoma; Adult Epithelioid Sarcoma; Adult Extraskeletal Chondrosarcoma; Adult Extraskeletal Osteosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Fibrous Histiocytoma; Adult Malignant Hemangiopericytoma; Adult Malignant Mesenchymoma; Adult Neurofibrosarcoma; Adult Synovial Sarcoma; Childhood Alveolar Soft-part Sarcoma; Childhood Angiosarcoma; Childhood Epithelioid Sarcoma; Childhood Fibrosarcoma; Childhood Leiomyosarcoma; Childhood Liposarcoma; Childhood Malignant Mesenchymoma; Childhood Neurofibrosarcoma; Childhood Synovial Sarcoma; Dermatofibrosarcoma Protuberans; Metastatic Childhood Soft Tissue Sarcoma; Nonmetastatic Childhood Soft Tissue Sarcoma; Stage I Adult Soft Tissue Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Neurofibrosarcoma; Sarcoma, Synovial; Dermatofibrosarcoma | interventions — Doxorubicin; Watchful Waiting; Observation; Radiotherapy, Conformal; Ifosfamide; indolepropanol phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A: No adjuvant treatment (Experimental): Patients with low-grade tumor with either negative or positive microscopic margins or high-grade tumor ≤ 5 cm (in maximum diameter) with negative microscopic margins are assigned to arm A: (observation only).
  Interventions: Other: clinical observation; Procedure: therapeutic conventional surgery
- Arm B: Low risk; adjuvant radiotherapy (Experimental): Patients with high-grade tumor ≤ 5 cm (in maximum diameter) with positive microscopic margins are assigned to arm B: (adjuvant radiotherapy). Beginning between 6-42 days after surgical resection, patients undergo a total of 31 fractions of adjuvant radiotherapy.
  Interventions: Other: clinical observation; Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy
- Arm C: Intermediate & High risk; adjuvant chemoradiotherapy (Experimental): High risk [metastatic, resected, incompletely resected, or unresected disease] patients with high-grade, grossly resected primary tumor, with metastases are assigned to receive arm C: (adjuvant chemoradiotherapy). Patients receive ifosfamide IV; doxorubicin hydrochloride IV; beginning in week 4, patients also undergo a total of 31 fractions of radiotherapy.
  Interventions: Drug: doxorubicin hydrochloride; Other: clinical observation; Radiation: 3-dimensional conformal radiation therapy; Drug: ifosfamide
- Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy (Experimental): High risk [metastatic, resected, incompletely resected, or unresected disease] patients with unresected, high-grade metastatic tumor are assigned to receive treatment as in arm D: (neoadjuvant chemoradiotherapy, surgery, and adjuvant chemotherapy with or without radiotherapy): Patients receive ifosfamide IV; doxorubicin hydrochloride IV. Beginning in week 4, patients also undergo a total of 31 fractions of radiotherapy. Patients undergo surgical resection in week 13.
  Interventions: Drug: doxorubicin hydrochloride; Other: clinical observation; Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy; Drug: ifosfamide

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
  Arms: Arm C: Intermediate & High risk; adjuvant chemoradiotherapy; Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy
Other: clinical observation — Patients undergo observation
  Other Names: observation
Procedure: therapeutic conventional surgery — Patients undergo surgery
  Arms: Arm A: No adjuvant treatment; Arm B: Low risk; adjuvant radiotherapy; Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy
Radiation: 3-dimensional conformal radiation therapy — Patients undergo radiotherapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
  Arms: Arm B: Low risk; adjuvant radiotherapy; Arm C: Intermediate & High risk; adjuvant chemoradiotherapy; Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
  Arms: Arm C: Intermediate & High risk; adjuvant chemoradiotherapy; Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy

SUMMARY:
This phase III trial is studying observation to see how well a risk based treatment strategy works in patients with soft tissue sarcoma. In the study, patients are assigned to receive surgery +/- radiotherapy +/- chemotherapy depending on their risk of recurrence. Sometimes, after surgery, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as ifosfamide and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define a risk-based treatment strategy comprising observation only, adjuvant radiotherapy, or adjuvant chemoradiotherapy or neoadjuvant chemoradiotherapy, surgery, and adjuvant chemotherapy with or without radiotherapy in young patients with non-rhabdomyosarcoma soft tissue sarcoma (NRSTS).

II. Assess event-free and overall survival of patients treated with these regimens.

III. Assess the pattern of treatment failure in these patients.

SECONDARY OBJECTIVES:

I. Assess the feasibility of a neoadjuvant chemoradiotherapy approach in patients with intermediate- or high-risk NRSTS.

II. Assess the imaging and pathologic responses to neoadjuvant chemoradiotherapy in patients with intermediate- or high-risk NRSTS.

III. Correlate imaging and pathologic response with clinical outcomes in patients with intermediate- or high-risk disease who undergo neoadjuvant chemoradiotherapy.

IV. Prospectively define clinical prognostic factors associated with event-free survival, overall survival, local recurrence, and distant recurrence in these patients.

V. Correlate patient outcomes with findings of biologic studies performed on tissue specimens collected on protocol COG-D9902 from these patients.

VI. Determine whether the diagnosis and histologic grade of NRSTS assigned by the enrolling institution correlates with the diagnosis and histologic grade established by central expert pathology reviewers.

VII. Compare the Pediatric Oncology Group (POG) and Fédération Nationale des Centres de Lutte Contre le Cancer (French Federation of Cancer Centers [FNCLCC]) pathologic grading systems to determine which better correlates with clinical outcomes.

OUTLINE: This is a multicenter study. Patients are divided into 3 risk groups according to presence of metastatic disease (yes vs no), status of prior surgery (resected vs unresected), grade of tumor (low vs high), and size of primary tumor (≤ 5 cm vs > 5 cm). Patients are assigned to different treatment regimens based on disease extent (nonmetastatic vs metastatic), tumor size (≤ 5 cm vs > 5 cm), extent of resection of primary tumor (resected vs unresected), extent of resection of metastases (complete or microscopic residual vs gross residual), microscopic tumor margins (negative vs positive), and tumor grade (low vs high).

GROUP 1 (low risk [nonmetastatic, grossly resected disease, except high-grade tumor > 5 cm]): Patients with low-grade tumor with either negative or positive microscopic margins or high-grade tumor ≤ 5 cm (in maximum diameter) with negative microscopic margins are assigned to regimen A. Patients with high-grade tumor ≤ 5 cm (in maximum diameter) with positive microscopic margins are assigned to regimen B.

REGIMEN A (observation only): Patients undergo observation only.

REGIMEN B (adjuvant radiotherapy): Beginning between 6-42 days after surgical resection, patients undergo a total of 31 fractions of adjuvant radiotherapy.

GROUP 2 (intermediate risk [nonmetastatic, resected or unresected disease]): Patients with grossly resected, high-grade tumor > 5 cm (in maximum diameter) are assigned to regimen C. Patients with unresected tumor are assigned to regimen D.

REGIMEN C (adjuvant chemoradiotherapy): Patients receive ifosfamide IV over 3 hours on days 1-3 in weeks 1, 4, 7, 10, 13, and 16 and doxorubicin hydrochloride IV over 24 hours on days 1 and 2 in weeks 1, 4, 13, 16, and 19. Beginning in week 4, patients also undergo a total of 31 fractions of radiotherapy.

*NOTE: *Patients who receive brachytherapy will initiate radiotherapy in Week 1. If brachytherapy is administered, chemotherapy should begin within 2 weeks of completion of brachytherapy and the Weeks 1 and 19 doxorubicin should be given instead at Weeks 7 and 10.

REGIMEN D (neoadjuvant chemoradiotherapy, surgery, and adjuvant chemotherapy with or without radiotherapy): Neoadjuvant chemoradiotherapy and surgery: Patients receive ifosfamide IV over 3 hours on days 1-3 in weeks 1, 4, 7, and 10 and doxorubicin hydrochloride IV over 24 hours on days 1 and 2 in weeks 1 and 4. Beginning in week 4, patients also undergo a total of 31 fractions of radiotherapy**. Patients undergo surgical resection in week 13.

NOTE: **Patients with primary hepatic tumors do not receive radiotherapy in week 4.

Adjuvant chemotherapy with or without radiotherapy: Patients receive ifosfamide IV over 3 hours on days 1-3 in weeks 16 and 19 and doxorubicin hydrochloride IV over 24 hours on days 1 and 2 in weeks 16, 19***, and 22. Beginning in week 16, patients achieving gross total resection with positive microscopic margins undergo a total of 6 fractions of adjuvant radiotherapy. Patients achieving less than total gross resection undergo a total of 11 fractions of adjuvant radiotherapy. Patients achieving total gross resection with negative microscopic margins do not receive adjuvant radiotherapy.

NOTE: ***Patients who receive adjuvant radiotherapy in week 16 receive doxorubicin hydrochloride in week 25 instead of week 19.

GROUP 3 (high risk [metastatic, resected, incompletely resected, or unresected disease]): Patients with low-grade, all-sites resected tumor with either negative or positive microscopic margins are assigned to receive treatment as in group 1 regimen A. Patients with high-grade, grossly resected primary tumor, and metastatic disease are assigned to receive treatment as in group 2 regimen C. Patients with unresected, high-grade metastatic tumor are assigned to receive treatment as in group 2 regimen D.

In all groups, treatment continues in the absence of disease progression. After completing study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-rhabdomyosarcoma soft tissue sarcoma (STS), confirmed by central pathology review via concurrent enrollment on protocol COG-D9902

  * Metastatic or non metastatic disease
* Meets 1 of the following criteria:

  * Intermediate (i.e., rarely metastasizing) or malignant STS, including any of the following:

    * Adipocytic tumor, including liposarcoma of any of the following histology subtypes:

      * Dedifferentiated
      * Myxoid
      * Round cell
      * Pleomorphic type
      * Mixed-type
      * Not otherwise specified (NOS)
    * Fibroblastic/myofibroblastic tumors, including any of the following:

      * Solitary fibrous tumor
      * Hemangiopericytoma
      * Low-grade myofibroblastic sarcoma
      * Myxoinflammatory fibroblastic sarcoma
      * Adult fibrosarcoma*
      * Myxofibrosarcoma
      * Low-grade fibromyxoid sarcoma or hyalinizing spindle-cell tumor
      * Sclerosing epithelioid fibrosarcoma
    * So-called fibrohistiocytic tumors, including any of the following:

      * Plexiform fibrohistiocytic tumor
      * Giant cell tumor of soft tissues
      * Pleomorphic malignant fibrous histiocytoma (MFH)/undifferentiated pleomorphic sarcoma
      * Giant cell MFH/undifferentiated pleomorphic sarcoma with giant cells
      * Inflammatory MFH/undifferentiated pleomorphic sarcoma with prominent inflammation
    * Smooth muscle tumor (leiomyosarcoma)
    * Pericytic [perivascular] tumor (malignant glomus tumor or glomangiosarcoma)
    * Vascular tumor, including angiosarcoma
    * Chondro-osseous tumors of any of the following types:

      * Mesenchymal chondrosarcoma
      * Extraskeletal osteosarcoma
    * Tumors of uncertain differentiation, including any of the following:

      * Angiomatoid fibrous histiocytoma
      * Ossifying fibromyxoid tumor
      * Myoepithelioma/parachordoma
      * Synovial sarcoma
      * Epithelioid sarcoma
      * Alveolar soft-part sarcoma
      * Clear cell sarcoma of soft tissue
      * Extraskeletal myxoid chondrosarcoma ("chordoid type")
      * Malignant mesenchymoma
      * Neoplasms with perivascular epithelioid cell differentiation (PEComa)
      * Clear cell myomelanocytic tumor
      * Intimal sarcoma
  * Malignant peripheral nerve sheath tumor
  * Dermatofibrosarcoma protuberans meeting both of the following criteria:

    * Non metastatic disease
    * Tumor must be grossly resected prior to study enrollment
  * Embryonal sarcoma of the liver
  * Unclassified STS that is too undifferentiated to be placed in a specific pathologic category (undifferentiated STS or STS NOS)
* Gross resection of the primary tumor ≤ 42 days prior to enrollment required except if any of the following circumstances apply:

  * Non metastatic high-grade tumor > 5 cm in maximal diameter and gross or microscopic residual tumor is anticipated after resection
  * Tumor of either high- or- low-grade that cannot be grossly excised without unacceptable morbidity
  * High-grade tumor with metastases

    * Patients with metastatic low-grade tumor whose disease is amenable to gross resection at all sites must undergo gross resection of all sites prior to study entry
* Patients with a tumor recurrence after a gross total resection are not eligible
* Tumors arising in bone are not eligible
* Patients with epithelioid sarcoma, clear cell sarcoma, or clinical or radiologic evidence of regional lymph node enlargement must undergo sentinel lymph node biopsies or lymph node sampling to confirm the status of regional lymph nodes* NOTE: *Except in cases where the study radiologist reviews the imaging and indicates that a biopsy is not needed to confirm that the patient has lymph node involvement.

  * If lymph node biopsies are positive for tumor (or the lymph nodes are classified as positive by the study radiologist), formal lymph node dissection must be done at the time of definitive surgery(prior to study entry for patients assigned to study regimen C)
* Patients with metastatic disease must undergo a biopsy to confirm the presence of metastatic tumor if all metastases are < 1 cm in maximal diameter (except in cases where the study radiologist reviews the imaging and indicated that a biopsy is not needed to confirm that the patient has metastatic disease)
* Lansky performance status (PS) 50-100% (for patients ≤ 16 years of age) OR Karnofsky PS 50-100% (for patients > 16 years of age)
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,000/mm³*
* Platelet count ≥ 100,000/mm³*
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min (≥ 40 mL/min for infants < 1 year of age)* or serum creatinine based on age and/or gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 year to < 2 years of age)
  * 0.8 mg/dL (2 years to < 6 years of age)
  * 1.0 mg/dL (6 years to < 10 years of age)
  * 1.2 mg/dL (10 years to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 years to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Patients with urinary tract obstruction by tumor must meet the renal function criteria listed above AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)*
* Shortening fraction ≥ 27% by echocardiogram* OR ejection fraction ≥ 50% by radionuclide angiogram*
* Not pregnant or nursing (patients undergoing radiotherapy and/or chemotherapy)

  * No nursing for ≥ 1 month after completion of study treatment in study regimens C or D
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* Negative pregnancy test
* No evidence of dyspnea at rest*
* No exercise intolerance*
* Resting pulse oximetry reading > 94% on room air (for patients with respiratory symptoms)*
* Prior treatment for cancer allowed provided the patient meet the prior therapy requirements
* No prior anthracycline (e.g., doxorubicin or daunorubicin) or ifosfamide chemotherapy for patients enrolled on arm C or arm D
* No prior radiotherapy to tumor-involved sites

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 588 (Actual)
Dates: Start 2007-02-05 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Spunt, MD, Principal Investigator — Children's Oncology Group
Locations (187):
- United States (165):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Oncology Group, Arcadia, California
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Nemours Childrens Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri-Columbia, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Hospital Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Derived] Crane JN, Xue W, Qumseya A, Barkauskas DA, Chau K, Tan SY, Hiniker S, Dasgupta R, Venkatramani R, Spunt SL, Weiss AR, Laetsch TW. Malignant peripheral nerve sheath tumors: a report from children's oncology group study ARST0332. J Natl Cancer Inst. 2025 Dec 12:djaf359. doi: 10.1093/jnci/djaf359. Online ahead of print. PMID 41386267
- [Derived] Alvarez E, He J, Spunt SL, Hayes-Jordan A, Kao SC, Parham DM, Million L, Weiss AR, Barkauskas DA. Lymph node metastases in paediatric and young adult patients with non-rhabdomyosarcoma soft tissue sarcoma (NRSTS): Findings from Children's Oncology Group (COG) study ARST0332. Eur J Cancer. 2023 Feb;180:89-98. doi: 10.1016/j.ejca.2022.11.014. Epub 2022 Nov 25. PMID 36566574
- [Derived] Venkatramani R, Xue W, Randall RL, Wolden S, Anderson J, Lopez-Terrada D, Black J, Kao SC, Shulkin B, Ostrenga A, Pappo A, Spunt SL. Synovial Sarcoma in Children, Adolescents, and Young Adults: A Report From the Children's Oncology Group ARST0332 Study. J Clin Oncol. 2021 Dec 10;39(35):3927-3937. doi: 10.1200/JCO.21.01628. Epub 2021 Oct 8. PMID 34623899
- [Derived] Million L, Hayes-Jordan A, Chi YY, Donaldson SS, Wolden S, Morris C, Terezakis S, Laurie F, Morano K, Fitzgerald TJ, Yock TI, Rodeberg DA, Anderson JR, Speights RA, Black JO, Coffin C, McCarville MB, Kao SC, Hawkins DS, Spunt SL, Randall RL. Local Control For High-Grade Nonrhabdomyosarcoma Soft Tissue Sarcoma Assigned to Radiation Therapy on ARST0332: A Report From the Childrens Oncology Group. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):821-830. doi: 10.1016/j.ijrobp.2021.01.051. Epub 2021 Feb 3. PMID 33548339
- [Derived] Spunt SL, Million L, Chi YY, Anderson J, Tian J, Hibbitts E, Coffin C, McCarville MB, Randall RL, Parham DM, Black JO, Kao SC, Hayes-Jordan A, Wolden S, Laurie F, Speights R, Kawashima E, Skapek SX, Meyer W, Pappo AS, Hawkins DS. A risk-based treatment strategy for non-rhabdomyosarcoma soft-tissue sarcomas in patients younger than 30 years (ARST0332): a Children's Oncology Group prospective study. Lancet Oncol. 2020 Jan;21(1):145-161. doi: 10.1016/S1470-2045(19)30672-2. Epub 2019 Nov 27. PMID 31786124
- [Derived] Spunt SL, Francotte N, De Salvo GL, Chi YY, Zanetti I, Hayes-Jordan A, Kao SC, Orbach D, Brennan B, Weiss AR, van Noesel MM, Million L, Alaggio R, Parham DM, Kelsey A, Randall RL, McCarville MB, Bisogno G, Hawkins DS, Ferrari A. Clinical features and outcomes of young patients with epithelioid sarcoma: an analysis from the Children's Oncology Group and the European paediatric soft tissue Sarcoma Study Group prospective clinical trials. Eur J Cancer. 2019 May;112:98-106. doi: 10.1016/j.ejca.2019.02.001. Epub 2019 Apr 5. PMID 30954717
- [Derived] Ferrari A, Chi YY, De Salvo GL, Orbach D, Brennan B, Randall RL, McCarville MB, Black JO, Alaggio R, Hawkins DS, Bisogno G, Spunt SL. Surgery alone is sufficient therapy for children and adolescents with low-risk synovial sarcoma: A joint analysis from the European paediatric soft tissue sarcoma Study Group and the Children's Oncology Group. Eur J Cancer. 2017 Jun;78:1-6. doi: 10.1016/j.ejca.2017.03.003. Epub 2017 Apr 7. PMID 28391003
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: No Adjuvant Treatment | Arm B: Low Risk; Adjuvant Radiotherapy | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy
Started | 222 | 21 | 122 | 223
Completed | 205 | 14 | 96 | 117
Not Completed | 17 | 7 | 26 | 106
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 7 | 25
Not completed — Physician Decision | 0 | 1 | 2 | 27
Not completed — Protocol Violation | 6 | 2 | 10 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Ineligible | 11 | 2 | 2 | 23
Not completed — Refusal of further protocol therapy | 0 | 1 | 3 | 15
Not completed — Inability to start week 16 tx on time | 0 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: No Adjuvant Treatment | Arm B: Low Risk; Adjuvant Radiotherapy | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy | Total
Number analyzed (Participants) | 222 | 21 | 122 | 223 | 588
Age, Continuous [Mean (Standard Deviation); unit: Months] | 138.87 (60.88) | 142.58 (59.46) | 155.14 (69.20) | 171.31 (68.90) | 154.68 (67.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 9 | 60 | 120 | 313
  Male | 98 | 12 | 62 | 103 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 1 | 22 | 38 | 90
  Not Hispanic or Latino | 185 | 19 | 95 | 178 | 477
  Unknown or Not Reported | 8 | 1 | 5 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3 | 6
  Asian | 7 | 1 | 2 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 23 | 2 | 21 | 43 | 89
  White | 169 | 16 | 90 | 137 | 412
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 22 | 2 | 7 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Probability for Event Free Survival.
Description: Probability of no relapse, secondary malignancy or death after 5 years since enrollment.
Time Frame: 5 years
Population: Ineligible patients are excluded as well as patients who were treated on the incorrect arm.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 5 years
Arm/Group | Arm A: No Adjuvant Treatment | Arm B: Low Risk; Adjuvant Radiotherapy | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy
Number analyzed (Participants) | 205 | 17 | 110 | 196
Probability of EFS at 5 years | 0.8984 [0.8395 to 0.9572] | 0.7647 [0.5348 to 0.9946] | 0.6079 [0.4818 to 0.7341] | 0.4873 [0.3951 to 0.5796]

2. Secondary Outcome: Toxicity Rate
Description: Percentage of Arm D patients experiencing grade 4+ adverse events.
Time Frame: 13 weeks
Population: Excluding ineligible patients and patients not treated based on the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm D: Intermediate & High Risk; Neoadjuvant chemoradiotherapy
Arm/Group | Arm D
Number analyzed (Participants) | 196
percentage of participants | 3.06 [0.65 to 5.47]

3. Secondary Outcome: Complete or Partial Response Rate
Description: Tumor response by imaging. Complete Response (CR): Complete disappearance of the tumor. Partial Response (PR): At least 64% decrease in volume compared to the measurement obtained at study enrollment. Overall Response (OR)=CR+PR.
Time Frame: 13 weeks
Population: Only Arm D patients were evaluated for imaging response at week 13 after surgery. Ineligible and inevaluable Arm D patients were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm D
Number analyzed (Participants) | 142
percentage of patients | 33.1 [25.36 to 40.84]

4. Secondary Outcome: Percent Tumor Necrosis
Description: Percent tumor necrosis by pathology review.
Time Frame: 13 weeks
Population: Only Arm D patients were evaluated at week 13 for percent tumor necrosis. Ineligible and inevaluable Arm D patients were excluded.
Measure: Mean (Standard Deviation); unit: percentage of tumor necrosis
Arm/Group | Arm D
Number analyzed (Participants) | 129
percentage of tumor necrosis | 59.4 (38.5)

5. Secondary Outcome: Event Free Survival Probability Disease Extent
Description: Probability of no relapse, secondary malignancy or death after 5 years since enrollment.
Time Frame: 5 years
Population: 94 participants were excluded because of ineligibility, incorrect treatment, or absence of evaluation for tumor invasiveness and histologic grade.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Non-metastatic | Metastatic
Number analyzed (Participants) | 425 | 69
Probability | 0.7758 [0.7202 to 0.8313] | 0.1960 [0.0742 to 0.3178]
Statistical Analysis 1: Comparison: Non-metastatic vs Metastatic; The Cox proportional hazards model was used to evaluate prognostic impact of disease extent (non-metastatic; metastatic) after accounting for the effects of site of the primary tumor (body wall; extremity; head/neck; visceral), tumor size (<=5cm; >5cm), tumor depth (deep; superficial), tumor invasiveness (invasive; non-invasive), extent of resection of the primary tumor (less than total resection; margin -; margin +), and histologic (POG) grade; Test type: Other; p < 0.0001, Regression, Cox

6. Secondary Outcome: Event Free Survival Probability Histologic Grade
Description: Probability of no relapse, secondary malignancy or death after 5 years since enrollment
Time Frame: 5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Histologic Grade 1 | Histologic Grade 2 | Histologic Grade 3
Number analyzed (Participants) | 60 | 79 | 355
Probability | 0.9636 [0.8943 to 1.0000] | 0.8505 [0.7382 to 0.9627] | 0.6136 [0.5442 to 0.6831]
Statistical Analysis 1: Comparison: Histologic Grade 1 vs Histologic Grade 2 vs Histologic Grade 3; The Cox proportional hazards model was used to evaluate prognostic impact of histologic (POG) grade after accounting for the effects of disease extent (non-metastatic; metastatic), site of the primary tumor (body wall; extremity; head/neck; visceral), tumor size (<=5cm; >5cm), tumor depth (deep; superficial), tumor invasiveness (invasive; non-invasive), and extent of resection of the primary tumor (less than total resection; margin -; margin +); Test type: Other; p = 0.0049, Regression, Cox

7. Secondary Outcome: Overall Survival Probability Disease Extent
Description: Probability of survival after 5 years since enrollment.
Time Frame: 5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Non-metastatic | Metastatic
Number analyzed (Participants) | 425 | 69
Probability | 0.8752 [0.8313 to 0.9190] | 0.3153 [0.1677 to 0.4629]
Statistical Analysis 1: Comparison: Non-metastatic vs Metastatic; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.0001, Regression, Cox

8. Secondary Outcome: Overall Survival Probability Extent of Resection of the Primary Tumor
Description: Probability of survival after 5 years since enrollment.
Time Frame: 5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Less Than Total Resection | Negative Margins | Positive Margins
Number analyzed (Participants) | 163 | 247 | 84
Probability | 0.5975 [0.4913 to 0.7036] | 0.9353 [0.8923 to 0.9782] | 0.7764 [0.6565 to 0.8963]
Statistical Analysis 1: Comparison: Less Than Total Resection vs Negative Margins vs Positive Margins; The Cox proportional hazards model was used to evaluate prognostic impact of the resection extent of the primary tumor (less than total resection; margin -; margin +) after accounting for the effects of site of the primary tumor (body wall; extremity; head/neck; visceral), disease extent (non-metastatic; metastatic), tumor size (<=5cm; >5cm), tumor depth (deep; superficial), tumor invasiveness (invasive; non-invasive), and histologic (POG) grade; Test type: Other; p = 0.0096, Regression, Cox

9. Secondary Outcome: Incidence of Distant Metastasis
Description: Percent of patients who had distant metastasis.
Time Frame: Up to 10 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-metastatic | Metastatic
Number analyzed (Participants) | 425 | 69
Percentage of participants | 10.59 [7.66 to 13.51] | 60.87 [49.35 to 72.39]
Statistical Analysis 1: Comparison: Non-metastatic vs Metastatic; The logistic regression model was used to evaluate prognostic impact of disease extent (non-metastatic; metastatic) after accounting for the effects of site of the primary tumor (body wall; extremity; head/neck; visceral), tumor size (<=5cm; >5cm), tumor depth (deep; superficial), tumor invasiveness (invasive; non-invasive), extent of resection of the primary tumor (less than total resection; margin -; margin +), and histologic (POG) grade; Test type: Other; p < 0.0001, Regression, Logistic; Firth logistic regression is used to overcome the issue of quasi-complete separation of data points

10. Secondary Outcome: Incidence of Distant Metastasis
Description: Percent of patients who had distant metastasis.
Time Frame: Up to 10 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Histologic Grade 1 | Histologic Grade 2 | Histologic Grade 3
Number analyzed (Participants) | 60 | 79 | 355
Percentage of participants | 0.00 [0.00 to NA] — Dispersion can't be estimated because no participants with histological grade 1 had a distant metastasis. | 5.06 [0.23 to 9.90] | 23.38 [18.98 to 27.78]
Statistical Analysis 1: Comparison: Histologic Grade 1 vs Histologic Grade 2 vs Histologic Grade 3; The logistic regression model was used to evaluate prognostic impact of histologic (POG) grade after accounting for the effects of disease extent (non-metastatic; metastatic), site of the primary tumor (body wall; extremity; head/neck; visceral), tumor size (<=5cm; >5cm), tumor depth (deep; superficial), tumor invasiveness (invasive; non-invasive), and extent of resection of the primary tumor (less than total resection; margin -; margin +); Test type: Other; p = 0.0228, Regression, Logistic; Firth logistic regression is used to overcome the issue of quasi-complete separation of data points

11. Secondary Outcome: Genetic and Gene Expression Profiles
Description: The tumors from patients registered on D9902 will be analyzed for genetic and gene expression profiles. The study will prospectively evaluate each tumor and confirm newly defined sarcoma diagnostic criteria based on cancer signatures in NRSTS.
Time Frame: At diagnosis
Population: None of the tumors were analyzed for genetic and gene expression profiles. The analysis will not be completed. The time frame "At diagnosis" is the time frame for the gene expression profiles.
Groups:
- All Patients: All patients
Arm/Group | All Patients
Number analyzed (Participants) | 0

12. Secondary Outcome: Degree of Agreement in Histologic Grade Determined by the Enrolling Institution Versus by Central Pathology Reviewers
Description: Histologic grades were determined by the central pathology reviewers and institutional pathologists based on published standards. A higher grade is associated with a more severe disease.
Time Frame: At Diagnosis
Population: Ineligible patients, as well as patients without histologic grade determined by enrolling institution or central pathology reviewers were excluded. The OM evaluates the degree of agreement of two pathology grading reviews at diagnosis. The time frame "At diagnosis" reflects the OM.
Measure: Number; unit: Participants
Arm/Group | Histologic Grade 1 by Enrolling Institution | Histologic Grade 2 by Enrolling Institution | Histologic Grade 3 by Enrolling Institution
Number analyzed (Participants) | 45 | 71 | 278
Participants
  Histologic grade 1 by central pathology reviewers | 38 | 5 | 1
  Histologic grade 2 by central pathology reviewers | 4 | 56 | 9
  Histologic grade 3 by central pathology reviewers | 3 | 10 | 268
Statistical Analysis 1: Comparison: Histologic Grade 1 by Enrolling Institution vs Histologic Grade 2 by Enrolling Institution vs Histologic Grade 3 by Enrolling Institution; Kappa statistic and its 95% confidence interval are used to assess agreement beyond random; Test type: Other; Kappa statistic = 0.82, 95% CI 2-sided [0.76 to 0.88]

13. Secondary Outcome: Degree of Agreement in Histologic Grade Between Pediatric Oncology Group (POG) and Fédération Nationale Des Centres de Lutte Contre le Cancer (FNCLCC) Pathologic Grading Systems
Description: POG and FNCLCC grades were determined by pathologists based on published standards. A higher grade is associated with a more severe disease.
Time Frame: At diagnosis
Population: Ineligible patients, as well as patients without histologic grade determined by POG or FNCLCC were excluded. The OM evaluates the degree of agreement of two pathology grading systems applied at diagnosis. The time frame "At diagnosis" reflects the OM.
Measure: Count of Participants; unit: Participants
Arm/Group | Histologic Grade 1 by FNCLCC | Histologic Grade 2 by FNCLCC | Histologic Grade 3 by FNCLCC
Number analyzed (Participants) | 79 | 222 | 241
Participants
  Histologic grade 1 by POG | 46 | 8 | 1
  Histologic grade 2 by POG | 24 | 69 | 0
  Histologic grade 3 by POG | 9 | 145 | 240
Statistical Analysis 1: Comparison: Histologic Grade 1 by FNCLCC vs Histologic Grade 2 by FNCLCC vs Histologic Grade 3 by FNCLCC; Kappa statistic and its 95% confidence interval are used to assess agreement beyond random; Test type: Other; Kappa statistic = 0.42, 95% CI 2-sided [0.36 to 0.48]

ADVERSE EVENTS:
Description: Ineligible patients and patients who were not treated based on the protocol were excluded from AE reporting (both serious and other).
Arm/Group | Arm A: No Adjuvant Treatment | Arm B: Low Risk; Adjuvant Radiotherapy | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy
Serious Adverse Events (participants affected / at risk) | 0/205 | 1/17 | 1/110 | 3/196
Other Adverse Events (participants affected / at risk) | 0/205 | 0/17 | 2/110 | 7/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: No Adjuvant Treatment (N=205) | Arm B: Low Risk; Adjuvant Radiotherapy (N=17) | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy (N=110) | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy (N=196)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: No Adjuvant Treatment (N=205) | Arm B: Low Risk; Adjuvant Radiotherapy (N=17) | Arm C: Intermediate & High Risk; Adjuvant Chemoradiotherapy (N=110) | Arm D: Intermediate & High Risk; Neoadjuvant Chemoradiotherapy (N=196)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.